CLINICAL TRIAL: NCT06770920
Title: Relief Of Airway Obstruction During Basic Life Support And Cardiopulmonary Resuscitation
Brief Title: Airway Obstruction During BLS
Acronym: BLS-OBST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université Paris-Sud (Other)
Responsible Party: Principal Investigator, Dan Benhamou, Study Principal Investigator, Université Paris-Sud
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: LabForSIMS 007
Record Dates: First submitted 2024-12-31; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Education Advancement
Keywords: simulation; education; observer tool; technical skills; basic life support

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- observer tool + (Experimental): use an observer tool
  Interventions: Other: use of an observer tool when not role-playing
- observer tool - (No Intervention): In this group, the students will not be given the observer tool and will observe other residents without any additional form.

INTERVENTIONS:
Other: use of an observer tool when not role-playing — Observers will use an observer tool (based on technical skills and specifically related to airway management during BLS) when they will be not role role-playing.
  Arms: observer tool +

SUMMARY:
Appropriate management of cardiac arrest (immediately and technically well performed) is a priority that must be taught to all citizens and future healthcare personnel, including future physicians. In this medical school, 2nd year medical students receive a 8 hour training session on basic life support (BLS) and management of cardiac arrest is taught into 5 successive parts, with learning and cumulative repetition of the steps: detection of unconsciousness, call for help, absence of breathing, cardiac massage and defibrillation.

During the many sessions previously carried out by our team, it often appeared that students, when evaluating breathing forget the 1st part related to airway and breathing, i.e. relieving airway obstruction. Yet it has been shown that opening the airway and early removal of a foreign body are associated with improved neurological survival. Importantly, mouth-to-mouth is not included in the learning session and compression-only is advocated.

The purpose of the present study is to evaluate if the use of an observation tool, with items centered on airway obstruction, can improve learning of this step, as shown in some previous trials.

This will be a trial performed in medical students in which training days will be randomized to include or not the use of an observation tool modified to emphasize the procedural parts that are aimed at relieving airway obstruction.

At the end of each day, students will be video-recorded while playing a short BLS scenario and airway obstruction-relieving skills will be compared.

DETAILED DESCRIPTION:
Appropriate management of cardiac arrest (immediately and technically well performed) is a priority that must be taught to all citizens and future healthcare personnel, including future physicians. In this medical school, 2nd year medical students receive a training session on basic life support (BLS) and management of cardiac arrest is taught into 5 successive steps, with learning and cumulative repetition of the steps: detection of unconsciousness, call for help, absence of breathing, cardiac massage and defibrillation.

During the many sessions previously carried out by our team, it often appeared that students, when evaluating breathing forget the 1st part related to airway and breathing, i.e. relieving airway obstruction. Yet it has been shown that opening the airway and early removal of a foreign body is associated with improved neurological survival. Importantly, mouth-to-mouth is not included in the learning session and compression-only is advocated.

The purpose of the present is to evaluate if the use of an observation tool, with items centered on airway obstruction, can improve learning of this step, as shown in some previous trials. In a previous trial indeed, the use of an observation tool improved airway management during simulated BLS but this was a secondary outcome and the validity of this result could not be ensured. To increase the positive effects of training when the learner is in the role of observer, some authors have proposed to strengthen the educational effect through the use of an observer tool that observers must complete by analyzing the progress of the task performed by their colleagues. This is a list describing a set of key points to be achieved. However, data concerning the educational value of these observer tools are limited. Studies on the use of these tools during crisis management training in the operating room assessed by high-fidelity simulation have shown improved learning outcomes although some other trials have provided negative results.

This will be a trial performed in medical students in which training days will be randomized to include or not the use of an observation tool modified to emphasize the procedural parts that are aimed at relieving airway obstruction.

This prospective and randomized study will be performed in an academic simulation center during a 8-hour basic emergency skills training in which life support during cardiac arrest lasts nearly 5 hours. Each of the 5 steps is taught incrementally and cumulatively (i.e. when an addition a step is taught, the next practical exercise starts from the 1st step and includes the new one), to familiarize students with technical skills and progression of care and to favor reflexivity by repetitively performing the task. For each step, the trainer initially evaluates the baseline knowledge of students, then provides theoretical information and finally all students perform the cumulative steps in dyads while being observed by the other trainees. The dyad strategy has been previously used and has been chosen to facilitate understanding of task distribution (call for help, lifting the chin during massage, defibrillator search and placement…) and improve training on how to change the rescuer performing the cardiac massage when fatigue arises.

Training days will be randomized according to the following design when learners will perform BLS:

* OT+ group: the observers will use an observer tool (based on technical skills and specifically highlighting actions related to airway management) when they will be not role role-playing. The OT will be provided to learners at the start of the session with a short briefing to explain how to use it. Sheets will be collected at the end of the session.
* OT- group: no observer tool will be used and observers will be encouraged to look at the performance of their peers.

The observer tool used will be based on the 2021 European Resuscitation Council Guidelines (amended when necessary with the 2023 ILCOR recommendations). The observer tool is made of 20 items but has been modified from a previous version to highlight the importance of airway obstruction by increasing the number of items related to airway management.

At the end of each day, students still working in randomly distributed dyads will be video-recorded while playing a short BLS scenario and airway relieving skills will be compared. Medical students will be enrolled after having given their written consent and video copyright. All scenarios will be recorded and anonymously retained and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* medical students participating in a full-day of basic life support training at the LabforSIMS- of Paris-Saclay medical school

Exclusion Criteria:

* declines active participation in the session
* no video-recording during simulation (i.e. technical problem)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-01-13 (Estimated); Primary Completion 2025-01-23 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
checklist describing performance of each dyad while performing BLS | From enrollment to the end of treatment at six months
  comparison of airway management skills, i.e. measured by external evaluation from the six items of the checklist related to this task between the OT + group and the OT- group among the checklist of items describing in detail the actions performed during BLS maximum score of 6/6 higher scores mean a better outcome Each item is scored 1 point

SECONDARY OUTCOMES:
checklist of the whole observer tool on task performance (20 items) | From enrollment to the end of treatment at six months
  Global performance of each dyad measured by external evaluation while performing BLS by comparing overall management skills, i.e. the 20 items between the OT + group and the OT- group maximum score of 20/20 higher scores mean a better outcome Each item is scored 1 point
Separate analysis of each of the 5 BLS sequences | From enrollment to the end of treatment at six months
  comparison of the performance of the two groups for each step of the checklist : detection of unconsciousness (4 items), call for help (4 items), absence of breathing (7 items), cardiac massage (5 items) and defibrillation (5 items). Each of the 5 steps is measured by external evaluation Each item is scored 1 point Higher scores indicate better performance
questionnaire satisfaction (post session) | From enrollment to the end of treatment at six months
  Satisfaction will be assessed by a Likert scale (0 to 10) (Kirkpatrick level 1
Questionnaire: educational value of an observer tool | From enrollment to the end of treatment at six months
  Perception about the educational value of an observer tool by a Likert scale (0 to 10) (Kirkpatrick level 1)
Multiple choice questions | From enrollment to the end of treatment at six months
  6 questions evaluating knowledge about BLS actions Maximum score 6 /6

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Goulamhoussen A, Havard C, Gille B, Francois B, Benhamou D, Blanie A. An observer tool to enhance learning of medical students during simulation training of cardiopulmonary resuscitation: a randomised controlled trial. BMC Med Educ. 2024 Jul 3;24(1):719. doi: 10.1186/s12909-024-05658-x. PMID 38961381
- [Result] Olasveengen TM, Semeraro F, Ristagno G, Castren M, Handley A, Kuzovlev A, Monsieurs KG, Raffay V, Smyth M, Soar J, Svavarsdottir H, Perkins GD. European Resuscitation Council Guidelines 2021: Basic Life Support. Resuscitation. 2021 Apr;161:98-114. doi: 10.1016/j.resuscitation.2021.02.009. Epub 2021 Mar 24. PMID 33773835
- [Result] Couper K, Abu Hassan A, Ohri V, Patterson E, Tang HT, Bingham R, Olasveengen T, Perkins GD; International Liaison Committee on Resuscitation Basic and Paediatric Life Support Task Force Collaborators. Removal of foreign body airway obstruction: A systematic review of interventions. Resuscitation. 2020 Nov;156:174-181. doi: 10.1016/j.resuscitation.2020.09.007. Epub 2020 Sep 16. PMID 32949674